CLINICAL TRIAL: NCT01408875
Title: Cardiac Rehabilitation and Low Frequency Electrical MyoStimulation in Chronic Heart Failure
Acronym: CREMS-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Gulf Estuarine Research Society (GERS) (Other); Bourgogne Association of Cardiology (Unknown); Ile-de-France Association of Cardiology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-03
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Cardiac rehabilitation; Exercise training; Peak VO2; Electrical myostimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation and EMS Group (Experimental): Patient Heart Failure who follows physical training and sessions of electrical quadricipital myostimulation.
  Interventions: Device: Low electrical myostimulation
- Rehabilitation Group only (No Intervention): Patient Heart Failure who follows physical training

INTERVENTIONS:
Device: Low electrical myostimulation — The group of patients randomized for additional EMS will have 20 sessions of 1 hour electrical quadricipital myostimulation.
  Arms: Rehabilitation and EMS Group

SUMMARY:
The purpose of this study is to determine if addition of low frequency electro-myo-stimulation to cardiac rehabilitation is effective to improve exercise capacity and/or muscular strength in chronic heart failure patients.

DETAILED DESCRIPTION:
In chronic heart failure, low exercise capacity is due, in part, to peripheral muscles abnormalities. Exercise training performed during cardiac rehabilitation improves exercise tolerance measured by cardiopulmonary exercise test. Low frequency electromyostimulation (EMS) was proposed as an alternative to exercise training (ET) in this population.

However, the effectiveness of the combination (EMS +ET) compared with ET alone is not proved. The main objective is to compare exercise capacity judged by peak VO2 after treatment by ET alone versus EMS+ET. The secondary end points are results on sub maximal parameters, muscular resistance, quality of life and effectiveness regarding clinical sub-groups.

This study is a controlled, randomized, multicentric (14 centres) designed to include 90 patients by group in two years period. Inclusion criteria are: CHF patients , NYHA class II to IIIb, with LVEF < 40% referred to complete a cardiac rehabilitation program.

All the patients benefit from a comprehensive cardiac rehabilitation program including educational program, therapeutical optimisation and exercise training for 20 sessions, 3 to 5 days a week. The group of patients randomized for additional EMS has 20 sessions of 1 hour electrical quadricipital myostimulation.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 75 yo
* stable Chronic Heart Failure (CHF) under "optimal" treatment since at least 1 week
* NYHA functional class II to IIIb
* left ventricular ejection fraction < 40%
* cardiopulmonary exercise test feasible
* whatever etiology of heart failure
* age of heart failure ≥ 3 months.
* have signed the consent document to participate in the study

Exclusion Criteria:

* previous treatment by functional electrical myo stimulation
* recent acute heart failure or inotropic intravenous agents used (< 10 days)
* recent coronary angioplasty (< 10 days)
* cardiac surgery < 1 month
* valvular disease requiring surgical treatment
* uncontrolled hypertension (≥ systolic 180 and/or diastolic 110 mmHg)
* severe respiratory insufficiency (VEMS < 1000 ml)
* pregnancy
* Automatic implantable defibrillator
* pace-makers : cardiac stimulation dependence or not known
* incapacity to achieve 6 min walk test and/or exercise testing
* absolute contra-indication to exercise test and/or exercise training
* myocarditis or pericarditis
* uncontrolled ventricular arrhythmias
* Obesity (BMI ≥ 35)
* known and documented peripheral myopathy
* participation to another study protocol
* patient incapable of giving consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Peak VO2 | at inclusion (baseline) then after 4 to 7 weeks of cardiac rehabilitation
  The primary outcome is the improvement of peak VO2 estimated by relative changes between before and at the end of the cardiac rehabilitation program.

SECONDARY OUTCOMES:
Changes on muscular strength | at inclusion then after 4 to 7 weeks of cardiac rehabilitation
  Measure of weight that the patient can lift 3 times but not four with quadriceps.
Changes on sub maximal parameters | at inclusion then after 4 to 7 weeks of cardiac rehabilitation
  Measure of ventilatory threshold and walk test of 6 min.
Modifications of quality of life | at inclusion then after 4 to 7 weeks of cardiac rehabilitation
  Minnesota questionnaire completed by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Marie Christine Iliou, MD, Principal Investigator — Hôpital Corentin Celton
Locations (14):
- France (14):
  - Centre de réadaptation spécialisé Saint Luc, Abreschviller
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Hospitalier de la Côte Fleurie, Cricquebœuf
  - Clinique SSR "Les Rosiers", Dijon
  - Hôpital Bocage Central, Dijon
  - Hôpital Corentin Celton, Issy-les-Moulineaux
  - Hôpital de Joigny, Joigny
  - Clinique de la Mitterie, Lomme
  - Centre Hospitalier Loire Vendée Ocean, Machecoul
  - Hôpital de jour de soins de suite et de réadaptation Léopold Bellan, Paris
  - Clinique Saint-Yves, Rennes
  - Hôpital Intercommunal Sud Léman Valserine, Saint-Julien-en-Genevois
  - Centre de réadaptation cardiaque Leopold Bellan, Tracy-le-Mont
  - Les Grands Prés, Villeneuve-Saint-Denis